CLINICAL TRIAL: NCT02339948
Title: A Phase II Trial of Stereotactic Body Radiation Therapy (SBRT) With or Without Intensity Modulated Radiation Therapy (IMRT) in the Treatment of Patients With Clinically Confined Prostate Adenocarcinoma
Brief Title: Phase II Trial of SBRT + or - IMRT in Treatment of Patients With Clinically Confined Prostate Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenesisCare USA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21C-2006-01
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Prostate Adenocarcinoma
Keywords: Locally confined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBRT only (Active Comparator): Patients assigned to this arm receive 8.0 Gy per fraction for 5 fractions for a total of 40 Gy
  Interventions: Radiation: SBRT
- IMRT plus SBRT Boost (Active Comparator): Patients assigned to this arm receive 1.8 Gy per fraction for 25 fractions over 5 weeks for a total of 45.0 Gy followed by an SBRT boost of 5.5 Gy per fraction for 4 fractions after IMRT for a total of 22.0 Gy
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — 8.0 Gy per fraction for 5 fractions for a total of 40 Gy
  Other Names: SBRT only

SUMMARY:
Patients with locally confined prostate adenocarcinoma (clinical stage T1c - T2bN0M0, Gleason score 7, PSA 20 ng/ml) are assigned to one of two treatment arms. Low risk patients (T1c-T2a and PSA <10 ng/ml and Gleason Score 6 or less) will receive 5 fractions of 8.0 Gy for a total of 40 Gy. Intermediate risk patients (T2b or PSA >10 ng/ml orGleason Score 7) will receive 1.8 Gy of IMRT for 25 fractions over 5 weeks for a total of 45 Gy. They will then receive a boost consisting of 4, 5.5 Gy fractions after IMRT for a total of 22 Gy.

DETAILED DESCRIPTION:
Patients with locally confined prostate adenocarcinoma (clinical stage T1c - T2bN0M0, Gleason score 7, PSA 20 ng/ml) are assigned to one of two treatment arms. Low risk patients (T1c-T2a and PSA <10 ng/ml and Gleason Score 6 or less) will receive 5 fractions of 8.0 Gy for a total of 40 Gy. Intermediate risk patients (T2b or PSA >10 ng/ml orGleason Score 7) will receive 1.8 Gy of IMRT for 25 fractions over 5 weeks for a total of 45 Gy. They will then receive a boost consisting of 4, 5.5 Gy fractions after IMRT for a total of 22 Gy. All patients will be assessed for toxicity at periodic time points following completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically determined adenocarcinoma is required.
* All other histologies are excluded.
* Tissue for diagnosis must be obtained by transrectal ultrasound biopsy.
* Gleason scoring classification of the biopsy specimen is required and must be greater than or equal to 7.
* 2002 AJCC clinical cancer stage as determined by either urologist or radiation oncologist must be T1c - T2b, N0, M0.
* N0 stage may be assigned following either negative imaging or negative pathologic assessment.
* Prostate volume as assessed by TRUS must be less than 60 cc. 3.1.5.
* PSA must be less than 20 ng/ml. ,
* Age ≥ 18,
* IPSS voiding symptoms score must be less than 18,
* Study consent form must be signed by the patient.

Exclusion Criteria:

* Gleason score of 8 - 10,
* Clinical stage T3 - T4,
* Age ≤ 18,
* Any evidence of nodal (N1) or distant (M1) disease,
* Prostate volume as assessed by TRUS > 60 cc,
* PSA > 20 ng/ml,
* IPSS voiding symptoms score > 18,
* Prior TURP,
* Prior pelvic radiotherapy or chemotherapy,
* Prior prostatectomy,
* Prior cancer other than basal cell or squamous cell skin carcinoma unless free of disease for > 5 years,
* Current medical or psychiatric illness that may interfere with treatment completion and followup,
* Hip prosthesis,
* Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2006-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of chronic grade 3 - 5 genitourinary (GU) and gastrointestinal (GI) toxicity of SBRT either as a boost following conventionally fractionated IMRT or as a monoradiotherapy | Periodical (baseline, during treatment, and at 1 month, 3 months, 6 months, 9 months, and 12 months post treatment. For the second and third years after therapy completion, follow-up visits will be every 6 months. Then annually for ____ years.
  At baseline, during treatment, and at 1 month, 3 months, 6 months, 9 months, and 12 months post treatment. For the second and third years after therapy completion, follow-up visits will be every 6 months. After the third year after therapy completion, follow-up visits will be annually for life, up to 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Mantz, MD, Principal Investigator — GenesisCare USA
Locations (4):
- United States (4):
  - 21st Century Oncology, Fort Myers, Florida
  - 21st Century Oncology, Plantation, Florida
  - 21st Century Oncology, Farmington Hills, Michigan
  - Century Oncology, Myrtle Beach, South Carolina